CLINICAL TRIAL: NCT02342743
Title: Open-trial on the Prevention of Chronic Migraines With the CEFALY Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cefaly Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 50207
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): Daily trigeminal nerve stimulation session of 20 minutes with CEFALY
  Interventions: Device: CEFALY

INTERVENTIONS:
Device: CEFALY

SUMMARY:
The main objective of this study was to assess the safety and efficacy of the Cefaly® e-TNS device as a prophylactic treatment of chronic migraine in adult patients.

DETAILED DESCRIPTION:
The purpose of this pilot study was to assess the safety and efficacy of the Cefaly® e-TNS device in the prophylactic treatment of chronic migraine in adult patients prior to implement a control trial where the size and final protocol will be specified thanks to the outcomes of this pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic migraine meeting the diagnostic criteria listed in ICHD-III beta (2013) section 1, migraine (1), with the exception of ''complicated migraine'' (i.e., hemiplegic migraine, migraine with brainstem aura, ophthalmoplegic migraine-recurrent painful ophthalmoplegic neuropathy, migrainous infarction) will be enrolled. They are required during baseline to have ≥15 headache days with each day consisting of ≥4 hours of continuous headache and with ≥50% of days being migraine or probable migraine days; and ≥4 distinct headache episodes, each lasting ≥4 hours.

Both patients with or without acute medication overuse (medication overuse headache - MOH) will be recruited

Exclusion Criteria:

1. Women: Pregnant, lactating or <6 months post partum
2. For patients already on treatment with medications in the following classes: antihypertensives, antidepressants, antiepileptics, no dose change of those medications is allowed for at least 3 months before start of baseline and during the entire study period.
3. For patients treated with Botox, no injection within 4 months before start of baseline or during the study.
4. Diagnosis of other primary or secondary headache disorders, except of Medication Overuse Headache
5. A Beck Depression Inventory score of >24 at baseline
6. Psychiatric disorders that could have interfered with study participation
7. Intolerance to supraorbital neurostimulation that makes the treatment not applicable (test of nociceptive threshold with specific Cefaly program)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Birlea, MD, Principal Investigator — Department of Neurology, University of Colorado Anschutz Medical Campus; Pierre Rigaux, Study Director — Cefaly Technology
Locations (1):
- University of Colorado Anschutz Medical Campus - Department of Neurology, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Daily trigeminal nerve stimulation session of 20 minutes with CEFALY
  CEFALY
Period: Baseline Period
Arm/Group | Active
Started | 73
Completed | 58
Not Completed | 15
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Change in prophylactic medication | 3
Not completed — Screening failure regarding baseline | 7
Period: Treatment Period
Arm/Group | Active
Started | 58 (7 patients didn't meet inclusion criteria for treatment period, evaluated at the end of the baseline)
Completed | 47
Not Completed | 11
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 8
Not completed — Change in prophylactic medication | 1

BASELINE CHARACTERISTICS:
Population: Participants who were included in the treatment period
Arm/Group | Active
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.45 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of headache episodes [Mean (Standard Deviation); unit: episodes] | 22.66 (5.35)
Number of headache days [Mean (Standard Deviation); unit: days] | 22.55 (5.38)
Number of moderate/severe headache days [Mean (Standard Deviation); unit: days] | 16.07 (7.65)
Number of migraine days [Mean (Standard Deviation); unit: days] | 19.02 (6.36)
Cumulative hours of headache on headache days [Mean (Standard Deviation); unit: hours] | 249.64 (124.29)
Average headache intensity [Mean (Standard Deviation); unit: units on a scale] — Headache intensity is defined on a scale from 0 (no pain) to 3 (maximum pain)
  units on a scale | 1.98 (0.44)
Acute medication use (total number) - all categories [Mean (Standard Deviation); unit: medications] | 26.33 (30.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Frequency of Headache Days
Description: Mean change in frequency of headache days (defined as a day with at least one headache episode, which is a patient-reported headache with pain) between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: days per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
days per 28-days | -3.12 (5.70)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change From Baseline in Acute Medication Intake
Description: Overall acute headache pain medication use (all categories) mean change between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: medications per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
medications per 28-days | -8.11 (18.74)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Frequency of Migraine Days
Description: Mean change in frequency of migraine days (any headache day is a migraine day, unless the pain intensity = 1 and there is no intake of acute anti-migraine medication) between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: days per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
days per 28-days | -3.35 (6.20)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Frequency of Moderate/Severe Headache Days
Description: Mean change in frequency of moderate/severe headache days (defined as a headache day with at least one headache episode with intensity = 2 or 3) between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: days per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
days per 28-days | -3.10 (5.98)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Monthly Cumulative Headache Hours
Description: Mean change in monthly cumulative headache hours on headache days between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: hours per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
hours per 28-days | -27.22 (80.46)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney) — Threshold for statistical significance set to 0.05

6. Secondary Outcome: Change in Frequency of Headache Episodes
Description: Mean change in frequency of headache episodes (defined as a patient-reported headache with pain) between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: episodes per 28-days
Arm/Group | Active
Number analyzed (Participants) | 58
episodes per 28-days | -3.12 (5.77)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: 50% Responder Rate for Migraine Days
Description: Number of subjects who observe a 50% reduction in the frequency of their migraine days between the 28-day baseline and the 28-day period ending with week 12 of treatment.
Time Frame: End of the 12 weeks treatment period
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 58
Participants | 11

8. Secondary Outcome: Change in the Average Headache Intensity
Description: Mean change in the average headache intensity between the 28-day baseline and the 28-day period ending with week 12 of treatment. Headache intensity is defined on a scale from 0 (no pain) to 3 (maximum pain).
Time Frame: End of baseline period and end of 12 weeks treatment period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 58
units on a scale | -0.12 (0.37)
Statistical Analysis 1: Comparison: Active; Test type: Superiority; p = 0.030, Wilcoxon (Mann-Whitney) — Threshold for statistical significance set to 0.05

ADVERSE EVENTS:
Time Frame: The AEs (adverse events) reported here were collected as of the first use of the device until the final visit after 12 weeks of stimulation
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 1/58
Other Adverse Events (participants affected / at risk) | 26/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=58)
Worsening myasthenia gravis and worsening migraine headache (Nervous system disorders) | 1 (1) — This SAE occurred the same day as the patient entered the treatment period but before using the Cefaly® device. Consequently, this SAE was considered not related to the use of the Cefaly® device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=58)
Cold, sinus infection, respiratory virus, sore throat, fever, flu-like symptoms (Infections and infestations) | 15 (21)
Gastroenteritis, stomach flu, norovirus (Infections and infestations) | 5 (7)
Vaginal infection (Infections and infestations) | 1 (1)
Migraine, worsening headaches (Nervous system disorders) | 5 (5)
Hives (Skin and subcutaneous tissue disorders) | 2 (2)
Surgical interventions (Surgical and medical procedures) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (3)
Skin irritation (Dermatitis forehead) (Skin and subcutaneous tissue disorders) | 1 (1) — Only these 2 AEs were related to the use of the Cefaly® device.
Burning sensation on forehead (Skin and subcutaneous tissue disorders) | 1 (1) — Only these 2 AEs were related to the use of the Cefaly® device.
Worsening vertigo (Nervous system disorders) | 1 (1)
Rash both arms and neck (Skin and subcutaneous tissue disorders) | 1 (1)
Kidney stone pain (Renal and urinary disorders) | 1 (1)
Diagnosis of fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 60 days from the time submitted to the sponsor for review. Sponsor may request:

* deletion of any trade secret, proprietary, or confidential information of Sponsor
* an additional 60 days to take measures to preserve its Intellectual Property rights

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT02342743/Prot_SAP_000.pdf